CLINICAL TRIAL: NCT00698932
Title: A 24-Week International, Multi-centre, Randomized, Parallel-group, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Saxagliptin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control With Diet and Exercise.
Brief Title: Evaluate Efficacy and Safety of Saxagliptin in Adult Patients With Type 2 Diabetes Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Peter Öhman, MD, PhD, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00005
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 inhibitors; HBA1c; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin 5mg (Experimental)
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — 5mg, oral tablet, once daily for 24 weeks
  Other Names: Onglyza
  Arms: Saxagliptin 5mg
Drug: Placebo — oral tablet, once daily for 24 weeks
  Arms: Placebo

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to evaluate the efficacy and safety in adult patients with inadequate glycaemic control with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes
* Patients should be drug naïve ie, not received medical treatment for diabetes,
* HbA1c ≥ 7.2% and ≤10.0% (at enrolment), HbA1c ≥ 7.0% and ≤10.0% (at randomization)

Exclusion Criteria:

* Insulin therapy within one year of enrolment (with the exception of insulin therapy during a hospitalization or use in gestational diabetes),
* Type 1 diabetes,history of ketoacidosis or hyperosmolar non-ketonic koma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Öhman, MD, PhD, Study Director — AstraZeneca, Wilmington, USA; Deborah Price, MSc, Study Chair — AstraZeneca, Wilmington, USA
Locations (30):
- China (15):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, China
  - Research Site, Chongqing, China
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Tianjin
- India (7):
  - Research Site, Hyderabaad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Coimbatore
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Makati City
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Quezon City
- South Korea (3):
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Daegu
  - Research Site, Seoul

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 5 mg: Saxagliptin 5 mg tablet, once daily (OD) for 24 weeks
- Placebo: Placebo tablet, once daily( OD) for 24 weeks
Period: Overall Study
Arm/Group | Saxagliptin 5 mg | Placebo
Started | 284 (Randomized and treated) | 284 (Randomized and treated)
Completed | 262 (Completed 24 Weeks of treatment) | 248 (Completed 24 Weeks of treatment)
Not Completed | 22 | 36
Not completed — Adverse Event | 0 | 2
Not completed — Incorrect enrollment | 0 | 2
Not completed — Study specific discontinuation criteria | 3 | 4
Not completed — Withdrawal by Subject | 11 | 23
Not completed — Lost to Follow-up | 6 | 1
Not completed — Severe non-compliance to protocol | 1 | 2
Not completed — Safety reasons | 0 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg | Placebo | Total
Number analyzed (Participants) | 284 | 284 | 568
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.23 (10.04) | 51.57 (10.34) | 51.4 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 129 | 253
  Male | 160 | 155 | 315

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 24 in Glycosylated Haemoglobin A1c (HbA1c)
Description: Adjusted* mean change from baseline in HbA1c achieved with saxagliptin 5 mg versus placebo at week 24 (LOCF, Full Analysis set). HbA1c is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. HbA1c data were excluded on and after rescue medication.
Time Frame: Baseline , Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis: change from baseline to Wk 24 LOCF for efficacy, subjects must have had a baseline and at least 1 post-baseline efficacy measurement. If participant received rescue medication, that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 277 | 274
percent
  Baseline | 8.15 (0.050) | 8.14 (0.050)
  Week 24 | 7.25 (0.063) | 7.75 (0.076)
  Adjusted Mean Change from Baseline | -0.84 (0.067) | -0.34 (0.065)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; *adjusted for baseline HbA1c; Mean Difference (Net) = -0.50, 95% CI [-0.65 to -0.34], Standard Error of Mean 0.079

2. Secondary Outcome: Absolute Change (mmol/L) From Baseline to Week 24 in Fasting Plasma Glucose (FPG)
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 5 mg versus placebo at week 24 (Last Observation Carried Forward (LOCF), Full Analysis set). FPG is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. FPG data were excluded on and after rescue medication.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 280 | 279
mmol/L
  Baseline | 9.15 (0.125) | 9.05 (0.141)
  week 24 | 8.10 (0.129) | 8.77 (0.163)
  Adjusted mean change from Baseline | -0.90 (0.144) | -0.17 (0.141)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; *adjusted for baseline FPG; Mean Difference (Net) = -0.73, 95% CI [-1.06 to -0.39], Standard Error of Mean 0.170

3. Secondary Outcome: Absolute Change (mg/dL) From Baseline to Week 24 in Fasting Plasma Glucose (FPG)
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 5 mg versus placebo at week 24 (LOCF, Full Analysis set). FPG is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. FPG data were excluded on and after rescue medication.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 280 | 279
mg/dL
  Baseline | 164.85 (2.253) | 163.03 (2.543)
  Week 24 | 145.97 (2.317) | 158.04 (2.942)
  Adjusted mean change from Baseline | -16.13 (2.586) | -3.01 (2.544)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; *adjusted for baseline FPG; Mean Difference (Net) = -13.12, 95% CI [-19.12 to -7.13], Standard Error of Mean 3.053

4. Secondary Outcome: Absolute Change (mmol*Min/L) From Baseline to Week 24 in Area Under the Curve (AUC) From 0 to 180 Minutes for Postprandial Glucose (PPG) During Mixed Meal (Instant Noodles) Tolerance Tests (MMTT) in All MMTT Participants
Description: Adjusted* mean change from baseline in PPG AUC achieved with saxagliptin 5 mg versus placebo at week 24 (LOCF, Full Analysis set). Trapezoidal method was used to compute AUC under the 3 hour PPG curve. Change from baseline for each subject is computed as the week 24 value minus the baseline value.PPG data were excluded on and after rescue medication
Time Frame: Baseline , Week 24
Population: MMTT was measured on a subset of patients in China cohort only at baseline and Wk 24. Randomized subjects, who took at least 1 dose of double-blind treatment to be included in analysis: change from baseline to Wk 24 (LOCF), must have had baseline and post-baseline data. Measurements observed on and after rescue medication were excluded.
Measure: Mean (Standard Error); unit: mmol*min/L
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 94 | 77
mmol*min/L
  Baseline | 2474 (46.9) | 2506 (64.9)
  Week 24 | 2063 (41.1) | 2262 (57.6)
  Adjusted mean change from Baseline | -417 (36.5) | -235 (40.4)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; *adjusted for baseline PPG AUC; Median Difference (Net) = -182, 95% CI [-289 to -74], Standard Error of Mean 54.4

5. Secondary Outcome: Absolute Change (mg*Min/dL) From Baseline to Week 24 in Area Under the Curve (AUC) From 0 to 180 Minutes for Postprandial Glucose (PPG) During Mixed Meal (Instant Noodles) Tolerance Tests (MMTT) in All MMTT Participants
Description: as for outcome 4
Time Frame: Baseline , Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 94 | 77
mg*min/dL
  Baseline | 44586 (844.8) | 45146 (1170.5)
  week 24 | 37166 (739.6) | 40751 (1036.6)
  Adjusted mean change from Baseline | -7534 (657.4) | -4255 (726.4)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; *adjusted for baseline PPG AUC; Mean Difference (Net) = -3280, 95% CI [-5214 to -1345], Standard Error of Mean 980.0

6. Secondary Outcome: Proportion of Patients Achieving a Therapeutic Glycemic Response Defined as HbA1c <7.0% at Week 24
Description: Proportion of participants (expressed in percentage of total participants) achieving HbA1c < 7.0% for saxagliptin versus placebo at week 24. HbA1c Data were excluded on and after rescue medication
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 277 | 274
Percentage of Participants | 45.8 | 28.8
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Net) = 17.0, 95% CI [8.9 to 24.9]

ADVERSE EVENTS:
Arm/Group | Saxagliptin 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/284 | 4/284
Other Adverse Events (participants affected / at risk) | 18/284 | 22/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg (N=284) | Placebo (N=284)
Angina Unstable (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Anal Injury (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Renal Abscess (Infections and infestations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg (N=284) | Placebo (N=284)
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator undertakes to provide AstraZeneca as soon as possible with preliminary data and drafts of proposed publications and disclosures, whether oral or in writing, and as soon as available, with the proposed final manuscript. AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed